CLINICAL TRIAL: NCT00277797
Title: A Randomized, Single-Blinded, Comparative Crossover Trial of the Safety and Efficacy of a Non-Invasive Targeted Electronic Pain Control Device ("Biowave System") Versus Transcutaneous Electrical Nerve Stimulation (TENS) for the Symptomatic Treatment of Chronic Low Back Pain.
Brief Title: Non-Invasive Targeted Electronic Pain Control Device ("Biowave System") Versus Transcutaneous Electrical Nerve Stimulation (TENS) for the Symptomatic Treatment of Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: BioWave Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 0102004819
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Low Back Pain
Keywords: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biowave first (Active Comparator): First Treatment: Biowave; Second Treatment: TENS
  Interventions: Device: Biowave Targeted Non-Invasive Electronic Pain Control Device; Device: TENS (Transcutaneous Electrical Nerve Stimulation) device
- TENS first (Active Comparator): First Treatment: TENS; Second Treatment: Biowave
  Interventions: Device: Biowave Targeted Non-Invasive Electronic Pain Control Device; Device: TENS (Transcutaneous Electrical Nerve Stimulation) device

INTERVENTIONS:
Device: Biowave Targeted Non-Invasive Electronic Pain Control Device — This device is a non-invasive non-pharmacologic treatment for pain. It sends a premixed modulated envelope of two high frequency electronic wave forms ("Feed Signals") between two electrodes.
  Other Names: Biowave
Device: TENS (Transcutaneous Electrical Nerve Stimulation) device — This device features a bisourced, biphasic waveform. The combined constant voltage, constant-current waveform provides a strong stimulus that allows the clinician to prescribe a treatment program.
  Other Names: Empi's (St. Paul, MN) Epix XL

SUMMARY:
Low back pain is a common condition, which extols a large cost to society from lost wages

The Biowave System was developed by Biowave Corporation (Biowave), Norwalk, CT. Two wires emanate from the unit. The feed wire is attached to a large disposable input pad ("Feed Electrode"). The return wire is attached to a smaller pad ("Return Electrode") over the source of the pain (the treatment site).

The device sends a premixed modulated envelope of two high frequency electronic wave forms ("Feed Signal") between the two electrodes. The beat frequency of the modulated envelope ("d-Frequency") is equal to the difference in frequency of the two feed signals. The location of beat frequency formation is dependent on the size and location of the two electrodes. With the configuration used in the study, the beat frequency signal is believed to form immediately ventrally to the Return electrode. The size of the volume of tissue affected can be changed and is dependent upon electrode geometry and the amplitude of the Feed Signal. The beat frequency is a low frequency blocking signal which is believed to cause a demodulation in the nerve cells and a reduction of the sodium/potassium ion exchange. As a result, the charge polarity of the nerve cell wall is prevented from changing and is therefore unable to transmit pain impulses. The size of the volume of tissue affected can be changed and is dependent upon electrode geometry and the amplitude of the Feed Signal.

The objective of this study is to compare the Biowave System with TENS (a currently available treatment) and to further evaluate its efficacy for the relief of pain in patients with chronic low back pain.

DETAILED DESCRIPTION:
Background-Low back pain is a common, costly & often chronic condition, estimated to affect 85% of people in their lifetime. A form of electronic pain control currently in use is TENS. Although the exact mechanism is not completely understood, it is proposed that its effectiveness is based on the gate control theory. Biowave has developed new patentable technology & a related device in the field of electromedicine. The device delivers a precise electrical signal to a specific volume of tissue in the body, which blocks the transmission of pain impulses.

Treatment Plan-Treatment will be initiated with device indicated by the order to which the pt. was randomized. Pts. will be connected to one of two devices hidden from view by application of two small round two-inch diameter electrodes to the lower back.

Baseline-A complete medical history & a physical examination will be performed. The pt. will complete a BPI questionnaire & be randomized to one of two treatment orders: 1) Biowave device followed by TENS device or 2) TENS device followed by Biowave Device. 2 treatment sessions will be separated by at least 72 hours.

Treatment-Prior to each treatment session, pt. will complete initial VAS evaluations. Pt.'s ROM will be assessed & vital signs will be obtained. Pts. will complete VAS & categorical pain assessments at end of the 20 minute treatment period.

Post-treatment-Pts. will repeat ROM test after device has been turned off & electrodes removed. VAS pain evaluations will be completed by the pt. at 30 & 60 minutes, vital signs & patient global impression of change will be obtained at 60 minutes following discontinuation of therapy. Pts. will be given VAS & categorical pain assessments to be completed at 4, 6, 12, 24 and 48 hours & 1 week after treatment (to be returned by mail/fax) to assess possible long-term analgesic effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be male or female of any race and between the ages of 18 and 60, inclusive;
* Female patients of childbearing potential may participate if they agree to a urine pregnancy test and the result is negative.
* The primary location of pain must be the lower back area (below 12th thoracic vertebra) without pain radiating to the legs (a subgroup [n=10] with pain radiating to the legs will be studied as well. Treatment will be initiated with the device indicated by the treatment order to which the patient was randomized). The pain must have been present for 3 months or greater prior to entry into the study;
* Patients must have a baseline score of ³40 mm on the VAS pain scale;
* If taking analgesics, patients must agree to maintain a steady regimen for the duration of the study;
* Patients must be able to understand and cooperate with study procedures; and
* Patients must have signed a legally effective written informed consent prior to entering the study.

Exclusion Criteria:

* Epilepsy
* Pregnancy
* Pacemaker
* History of cardiac arrhythmias
* Implantable devices (AICD, pump, etc.)
* Surgical intervention during the past month for the treatment of low back pain or its underlying etiology
* Other severe pain that may confound assessment or self-evaluation of the chronic low back pain;
* Patients with pending Worker's Compensation claims, pending civil litigation pertinent to the cause of low back pain, currently receiving monetary compensation for the injury resulting in back pain, or currently involved in out-of-court settlements for claims pertinent to their back pain;
* Abuse of illicit drugs or alcohol within the last 6 months;
* Clinically significant or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise participation in the study;
* Participation in a clinical trial for an investigational drug and/or agent within 30 days prior to screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2001-02; Primary Completion 2006-03 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Comparison of mean pain scores ("deep" pain and "superficial" or "surface" pain visual analog scales [VAS]) | determined at baseline, 20 minutes after optimization of signal amplitude, and at 30 and minutes 60 following discontinuation of treatm

SECONDARY OUTCOMES:
Range of motion test | before and after treatment
Patient global impressions of change (PGIC) | at end of treatment, and one day and one week after treatment
Mean pain scores to assess duration of analgesia. | at 4, 6, 12, 24 and 48 hours following discontinuation of treatment
Nature, frequency, and intensity of adverse events. | continuous
Physical examination and assessment of vital signs. | baseline, pre-treatment, and post-treatment
follow-up phone interviews. | one day and one week post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hugh C. Hemmings Jr., MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

REFERENCES:
- See also: Sponsor Website — http://www.biowave.com